CLINICAL TRIAL: NCT03102749
Title: Mechanism and Dynamics of Bronchial Hyper-reactivity to Methacholine in Distal Airway on Obese Patients With Asthma
Acronym: SCANN'AIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 8836; 2011-A01396-35 (Other: ANSM)
Record Dates: First submitted 2015-06-05; First posted 2017-04-06 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Airways; asthma; overweight
MeSH Terms: conditions — Asthma; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal weight: Included patients with a BMI < 25 will be part of this group.
  Interventions: Other: metacholine provocation test and CT-scan low dose
- Overweight: Included patients with a BMI >= 25 and <30 will be part of this group.
  Interventions: Other: metacholine provocation test and CT-scan low dose
- Obese: Included patients with a BMI >= 30 will be part of this group.
  Interventions: Other: metacholine provocation test and CT-scan low dose

INTERVENTIONS:
Other: metacholine provocation test and CT-scan low dose — Investigators perform a metacholine provocation test where expiratory CT slices were acquired at each dose

SUMMARY:
New insights of small airway contribution to asthma have been gained. Poor levels of control and recurrent exacerbations were shown to have the phenotypic counterpart of asthma with predominant small airway involvement. Very few pathological specificities were identified at this site: mast cells infiltration was suggested as the specific inflammatory change when compared to the proximal airways.Biomarkers in asthma are still complex to validate, especially in the blood, since compartmentalisation is intense in the lung and the airways, a property attributed to the filtering role of the lung to maintain homeostasis. Over the last few years, Fraction exhaled Nitric Oxide (FENO) was developed as a non-invasive and indirect reflection of airway eosinophilic inflammation]. In the blood, peripheral eosinophil counts were shown as a correct T helper 2 (TH2)-phenotype identifier but not perfectly related to airway eosinophilic infiltration. Club cell secretory protein (SCGB1A1) levels have been shown to have some relevance in asthma, chronic obstructive pulmonary disease (COPD), BOS, sarcoidosis, and lung cancer.A biomarker for small airway disease in asthma may improve the management of the disease, identify areas of therapeutic resistance and constitute a therapeutic guidance tool. In this study, investigators aimed to assess small airway involvement in asthmatic women as far as they could. For this purpose, investigators analysed trends in air trapping by acquiring expiratory CT slices at each dose during a bronchoprovocation test with metacholine. Biomarkers were subsequently tested and confronted to clinical and demographical characteristics in their ability to predict the small airway involvement index obtained at CT.

DETAILED DESCRIPTION:
Patients will be recruited in the respiratory department of University Hospital in Montpellier (France) from June 2012 to March 2014. All patients are asthmatics, in order to avoid any gender-related biases, investigators decided to include only women. All participants had normal range spirometry, specifically regarding forced expiratory volume. Each patient will undergo a bronchial provocation test coupled with a thoracic CT scan. Bronchial and alveolar Nitric Oxyde will also be measured, a blood sample will be obtained in order to measure biomarker concentrations, and the patients will be asked to answer the validated Asthma Control Questionnaire in order to quantify asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Female >= 18 yrs
* Asthma
* Treated with Inhaled Corticosteroid (ICS)
* normal range spirometry

Exclusion Criteria:

* Patients with other respiratory disease
* Patients with myocardial infarction (for 3 month before enrollment)
* Patients with cerebrovascular accident (for 3 month before enrollment)
* Patients with arterial aneurysm known
* Patients in pregnancy
* Patients nursing

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in the respiratory department of University Hospital in Montpellier (France) from June 2012 to March 2014. All patients are asthmatics, in order to avoid any gender-related biases, investigators decided to include only women. All participants had normal range spirometry, specifically regarding forced expiratory volume.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory:expiratory mean lung density | 4 hours (after the enrollment)
  Baseline versus post-methacholine challenge

SECONDARY OUTCOMES:
Change in lung fractal dimension | 4 hours (after the enrollment)
  Baseline versus post-methacholine challenge
Bronchial morphometry | Baseline
  Analysis of CT imaging
CC10 level | Baseline
  Clara cell 10 kD protein levels in blood
FeNO | Baseline
  Exhaled nitric oxide level
FaNO | Baseline
  Alveolar nitric oxide level

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud BOURDIN, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Department of respiratory disease, Montpellier, France

REFERENCES:
- See also: SCANN'AIR on the Open Science Framework — https://osf.io/acb84/
- See also: Derived methods publication. — https://doi.org/10.3389/fams.2019.00022
- See also: Secondary results publication. — https://www.ncbi.nlm.nih.gov/pubmed/?term=28108336